CLINICAL TRIAL: NCT03577912
Title: Efficacy of Transversus Abdominis Plane (TAP) Block Techniques: A Comparison Between Intraoperative Surgeon Administration by Direct Visualization vs Image Guided Administration by Anesthesiologist, a Prospective Randomized Controlled Trial
Brief Title: Efficacy of Transversus Abdominis Plane (TAP) Block Techniques: Surgeon vs Anesthesia - Ultrasound Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Cataldo, Instructor in Surgery, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P000347
Record Dates: First submitted 2018-06-25; First posted 2018-07-05 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Post Operative Analgesia; Non-inferiority Trial
Keywords: ERAS; transversus_abdominis_plane_block; postoperative_pain

STUDY DESIGN:
Intervention Model Description: prospective, randomized, patient and observer blinded non-inferiority trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patients, and all data collectors were blinded regarding which group the patients were in. Surgeons who performed the case were aware of the method used but were not involved with the data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block administered by Surgery (Active Comparator): transversus abdominis (TAP) plane block is performed by the surgeon at the conclusion of the surgery, still under general anesthesia, prior to removing the trocars a single dose 60 cc of 0.5%bupivicaine is delivered into the TAP under direct surgeon observed laparoscopic visualization. (Split dose 30cc/side)
  Interventions: Procedure: TAP block administered by Surgery
- TAP block administered by Anesthesia (Active Comparator): transversus abdominis (TAP) plane block is performed by the anesthesiologist at the conclusion of the surgery after incisions are closed and dressing are on, prior to emergence from general anesthesia, a single dose 60 cc of 0.5%bupivicaine is delivered into the TAP under by the anesthesiologist using ultrasound visualization. (Split dose 30cc/side)
  Interventions: Procedure: TAP block administered by Anesthesia

INTERVENTIONS:
Procedure: TAP block administered by Surgery — TAP block administered by Surgery
  Arms: TAP block administered by Surgery
Procedure: TAP block administered by Anesthesia — TAP block administered by Anesthesia
  Arms: TAP block administered by Anesthesia

SUMMARY:
The transversus abdominis plane (TAP) block is a regional anesthesia technique where local anesthetic is injected into the neurovascular plane between the transversus abdominis and internal oblique muscles. The TAP block has been shown to provide postoperative analgesia following abdominal surgery.There are many methods to administer local anesthetic into the transversus abdominus plane to provide post-operative analgesia. The more prevalent method is for an anesthesia provider to inject local anesthetic into the plane using ultrasound guidance, before surgery or after the conclusion of surgery. Alternatively, a surgeon can administer the local anesthetic during the operation without additional time or expense using direct laparoscopic visualization. We propose to compare the two methods for non-inferiority, in the context of an established enhanced recovery after surgery (ERAS) program. Non-inferiority being established by no demonstrable difference in post-operative narcotic requirements and equivalent average pain scores.

DETAILED DESCRIPTION:
Purpose: To demonstrate that TAP blockade administered by the surgeon during surgery is as effective as when placed as a separate procedure by an anesthesiologist under ultrasound guidance by head to head randomized comparison controlling for medication, concentration volume and location.

Introduction:

The transversus abdominis plane (TAP) block is a regional anesthesia technique where local anesthetic is injected into the neurovascular plane between the transversus abdominis and internal oblique muscles. The ventral rami of the segmental thoracolumbar nerves course through the TAP before innervating the anterolateral abdominal wall. The TAP block has been shown to provide postoperative analgesia following abdominal surgery. Prospective randomized trials have demonstrated analgesic efficacy of TAP block and cadaveric studies have shown reliable dye spread from T9-L1 (iliac crest to the costal margin) , although the spread is dependent upon the technique of injection, single versus multiple injections. The TAP block is an intermuscular plane block i.e., needle placed in the plane between the internal oblique and transversus abdominis muscles. The sensory fibers located in this plane is too small to be visualized by ultrasound or localized by nerve stimulation. The TAP block may be performed in patients under general anesthesia since nerve localization is not necessary. This block has a number of advantages which include technical simplicity, high analgesic effectiveness, opioid sparing, long duration of effect, up to 36 hours, minimal side effects in comparison to that associated with neuraxial analgesia (e.g., hypotension, motor blockade). TAP block has successfully been incorporated in enhanced recovery after surgery (ERAS) protocols to reduce postoperative pain, reduce post op narcotic requirement, provide earlier return of bowel function and reduce length of stay. However multiple techniques for placement of the block have been described, in differing locations and with differing agents to analgesia after a variety of procedures. Historically the block has been placed based on anatomic land marks in the triangle of Petit guided by the sensation of the administrator. The safety and anatomic reliability of this approach has been questioned. Currently the block is frequently placed by an anesthesiologist under ultrasound guidance. Recently there have been published reports of surgeons placing TAP blocks intraoperatively guided by palpation and direct visualization, both open and with laparoscopic visualization . It is currently the practice in the division of colon and rectal surgery to use a standardized method for placing a TAP block after open and laparoscopic abdominal colon and rectal cases as part of our ERAS protocol requiring minimal time and cost limited to the cost of the medication. The authors hypothesize that TAP block administered by the surgeon is as effective as when administered by an anesthesiologist under ultrasonic guidance controlling for medication, volume, concentration and location of placement.

Methods: This study is a randomized trial with a placebo control arm to confirm effectiveness of the block its self, as TAP block is fully adopted as standard practice throughout abdominal surgery. Consecutive patients 18 years old or greater with intellectual capacity to consent, who are scheduled to undergo elective open or laparoscopic abdominal surgery by the division of colorectal surgery, will be offered inclusion in the study. Choice of open versus laparoscopic procedure is at surgeons discretion based on the patient's condition, diagnosis and best practice. Those patients whose procedure begins laparoscopically who require conversion to laparotomy will be noted and included in the open group. Exclusions will include patients who have allergies to the medications, patients with a preoperative addiction to narcotics or chronic pain syndromes requiring chronic medication, or whose anatomy or procedure precludes placement of the block.

Consenting patients will be randomized to receive administration of a TAP block either intraoperatively by the surgeon by direct palpation and/or visualization or by an anesthesiologist under ultrasound guidance. Secondary randomization will assign 1/4rd of both arms to receive placebo. In treatment arm cases Marcaine 0.25% with epinephrine 1:200,000 in a volume in ccs equal to the patients weight in Kg will be delivered. Those assigned to placebo will receive an equivalent volume of saline. In all cases the block will be placed at the conclusion of the case; for the surgeon, prior to closure of the abdomen, for the anesthesiologist after skin closure but prior to emergence from general anesthesia.

The volume will be divided equally, bilaterally and injection via needle and syringe into the transversus abdominis muscle plane lateral to the border of the rectus muscle at the level of the umbilicus. In cases of longer xyphoid to pubis laparotomy incisions the volume of injection can be further divided to be injected superiorly and inferiorly in the abdominal wall to assure adequate distribution. In all cases the injection will be performed under general anesthesia after the completion of the case either immediately before closure of the abdominal incision(s) or immediately after closure, prior to emergence from anesthesia.

The patients and the data collection staff will be blinded at to the medication vs placebo and the method of administration.

Post operatively all patients in all groups will be included in a standard post-operative ERAS pathway including use of intravenous ketorolac and acetaminophen, metoclopramide, early ambulation. All patients will have access to standard post-operative analgesia including intravenous narcotics (morphine, hydromorphone) patient controlled analgesia (PCA) and PO analgesia acetaminophen, ibuprofen, oxycodone.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients undergoing laparoscopic colorectal resection in the division of colorectal surgery from March 2016 and April 2018 were eligible.
* Over 18 years old
* Intellect sufficient to sign consent, interpret analog pain scale

Exclusion Criteria:

* allergies to bupivacaine or epinephrine
* preoperative chronic narcotic usage
* chronic pain syndrome
* anatomy thought to preclude effective placement of the TAP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
narcotic requirement | first 48 hours after surgery
  overall narcotic medications used by the patient (in morphine equivalents)PACU, 6,12,25,and 48 hours after surgery
visual analogue pain scale - resting | first 48 hours after surgery
  visual analogue pain scale 0-10 observed at rest in the post-anesthesia care unit, 6,12,25,and 48 hours after surgery (0 = no pain, 10 = worst imaginable pain)
visual analogue pain scale - moving | first 48 hours after surgery
  visual analogue pain scale 0-10 observed with motion in post-anesthesia care unit, 6,12,25,and 48 hours after surgery (0 = no pain, 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Cataldo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Zhuang CL, Ye XZ, Zhang XD, Chen BC, Yu Z. Enhanced recovery after surgery programs versus traditional care for colorectal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2013 May;56(5):667-78. doi: 10.1097/DCR.0b013e3182812842. PMID 23575408
- [Background] Lee L, Mata J, Ghitulescu GA, Boutros M, Charlebois P, Stein B, Liberman AS, Fried GM, Morin N, Carli F, Latimer E, Feldman LS. Cost-effectiveness of Enhanced Recovery Versus Conventional Perioperative Management for Colorectal Surgery. Ann Surg. 2015 Dec;262(6):1026-33. doi: 10.1097/SLA.0000000000001019. PMID 25371130
- [Background] Carmichael JC, Keller DS, Baldini G, Bordeianou L, Weiss E, Lee L, Boutros M, McClane J, Feldman LS, Steele SR. Clinical Practice Guidelines for Enhanced Recovery After Colon and Rectal Surgery From the American Society of Colon and Rectal Surgeons and Society of American Gastrointestinal and Endoscopic Surgeons. Dis Colon Rectum. 2017 Aug;60(8):761-784. doi: 10.1097/DCR.0000000000000883. No abstract available. PMID 28682962
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Hain E, Maggiori L, Prost A la Denise J, Panis Y. Transversus abdominis plane (TAP) block in laparoscopic colorectal surgery improves postoperative pain management: a meta-analysis. Colorectal Dis. 2018 Apr;20(4):279-287. doi: 10.1111/codi.14037. PMID 29381824
- [Background] Johns N, O'Neill S, Ventham NT, Barron F, Brady RR, Daniel T. Clinical effectiveness of transversus abdominis plane (TAP) block in abdominal surgery: a systematic review and meta-analysis. Colorectal Dis. 2012 Oct;14(10):e635-42. doi: 10.1111/j.1463-1318.2012.03104.x. PMID 22632762
- [Background] Pirrera B, Alagna V, Lucchi A, Berti P, Gabbianelli C, Martorelli G, Mozzoni L, Ruggeri F, Ingardia A, Nardi G, Garulli G. Transversus abdominis plane (TAP) block versus thoracic epidural analgesia (TEA) in laparoscopic colon surgery in the ERAS program. Surg Endosc. 2018 Jan;32(1):376-382. doi: 10.1007/s00464-017-5686-7. Epub 2017 Jul 1. PMID 28667547
- [Background] Elkassabany N, Ahmed M, Malkowicz SB, Heitjan DF, Isserman JA, Ochroch EA. Comparison between the analgesic efficacy of transversus abdominis plane (TAP) block and placebo in open retropubic radical prostatectomy: a prospective, randomized, double-blinded study. J Clin Anesth. 2013 Sep;25(6):459-65. doi: 10.1016/j.jclinane.2013.04.009. Epub 2013 Aug 17. PMID 23965191
- [Background] Keller DS, Ermlich BO, Delaney CP. Demonstrating the benefits of transversus abdominis plane blocks on patient outcomes in laparoscopic colorectal surgery: review of 200 consecutive cases. J Am Coll Surg. 2014 Dec;219(6):1143-8. doi: 10.1016/j.jamcollsurg.2014.08.011. Epub 2014 Sep 16. PMID 25442068
- [Background] Gao T, Zhang JJ, Xi FC, Shi JL, Lu Y, Tan SJ, Yu WK. Evaluation of Transversus Abdominis Plane (TAP) Block in Hernia Surgery: A Meta-analysis. Clin J Pain. 2017 Apr;33(4):369-375. doi: 10.1097/AJP.0000000000000412. PMID 27518492
- [Background] Favuzza J, Delaney CP. Laparoscopic-guided transversus abdominis plane block for colorectal surgery. Dis Colon Rectum. 2013 Mar;56(3):389-91. doi: 10.1097/DCR.0b013e318280549b. PMID 23392158
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Park SY, Park JS, Choi GS, Kim HJ, Moon S, Yeo J. Comparison of Analgesic Efficacy of Laparoscope-Assisted and Ultrasound-Guided Transversus Abdominis Plane Block after Laparoscopic Colorectal Operation: A Randomized, Single-Blind, Non-Inferiority Trial. J Am Coll Surg. 2017 Sep;225(3):403-410. doi: 10.1016/j.jamcollsurg.2017.05.017. Epub 2017 Jun 10. PMID 28610880
- [Background] Fields AC, Gonzalez DO, Chin EH, Nguyen SQ, Zhang LP, Divino CM. Laparoscopic-Assisted Transversus Abdominis Plane Block for Postoperative Pain Control in Laparoscopic Ventral Hernia Repair: A Randomized Controlled Trial. J Am Coll Surg. 2015 Aug;221(2):462-9. doi: 10.1016/j.jamcollsurg.2015.04.007. Epub 2015 Apr 22. PMID 26206644
- [Background] Schumi J, Wittes JT. Through the looking glass: understanding non-inferiority. Trials. 2011 May 3;12:106. doi: 10.1186/1745-6215-12-106. PMID 21539749
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Ma N, Duncan JK, Scarfe AJ, Schuhmann S, Cameron AL. Clinical safety and effectiveness of transversus abdominis plane (TAP) block in post-operative analgesia: a systematic review and meta-analysis. J Anesth. 2017 Jun;31(3):432-452. doi: 10.1007/s00540-017-2323-5. Epub 2017 Mar 7. PMID 28271227
- [Background] Torgeson M, Kileny J, Pfeifer C, Narkiewicz L, Obi S. Conventional Epidural vs Transversus Abdominis Plane Block with Liposomal Bupivacaine: A Randomized Trial in Colorectal Surgery. J Am Coll Surg. 2018 Jul;227(1):78-83. doi: 10.1016/j.jamcollsurg.2018.04.021. Epub 2018 May 1. PMID 29723578
- [Background] Niraj G, Kelkar A, Hart E, Horst C, Malik D, Yeow C, Singh B, Chaudhri S. Comparison of analgesic efficacy of four-quadrant transversus abdominis plane (TAP) block and continuous posterior TAP analgesia with epidural analgesia in patients undergoing laparoscopic colorectal surgery: an open-label, randomised, non-inferiority trial. Anaesthesia. 2014 Apr;69(4):348-55. doi: 10.1111/anae.12546. PMID 24641640
- [Background] Barrington MJ, Ivanusic JJ, Rozen WM, Hebbard P. Spread of injectate after ultrasound-guided subcostal transversus abdominis plane block: a cadaveric study. Anaesthesia. 2009 Jul;64(7):745-50. doi: 10.1111/j.1365-2044.2009.05933.x. PMID 19624629
- [Background] Oh TK, Lee SJ, Do SH, Song IA. Transversus abdominis plane block using a short-acting local anesthetic for postoperative pain after laparoscopic colorectal surgery: a systematic review and meta-analysis. Surg Endosc. 2018 Feb;32(2):545-552. doi: 10.1007/s00464-017-5871-8. Epub 2017 Oct 26. PMID 29075970
- [Background] Rashid A, Gorissen KJ, Ris F, Gosselink MP, Shorthouse JR, Smith AD, Pandit JJ, Lindsey I, Crabtree NA. No benefit of ultrasound-guided transversus abdominis plane blocks over wound infiltration with local anaesthetic in elective laparoscopic colonic surgery: results of a double-blind randomized controlled trial. Colorectal Dis. 2017 Jul;19(7):681-689. doi: 10.1111/codi.13578. PMID 27943522
- [Background] Ventham NT, O'Neill S, Johns N, Brady RR, Fearon KC. Evaluation of novel local anesthetic wound infiltration techniques for postoperative pain following colorectal resection surgery: a meta-analysis. Dis Colon Rectum. 2014 Feb;57(2):237-50. doi: 10.1097/DCR.0000000000000006. PMID 24401887
- [Derived] Wong DJ, Curran T, Poylin VY, Cataldo TE. Surgeon-delivered laparoscopic transversus abdominis plane blocks are non-inferior to anesthesia-delivered ultrasound-guided transversus abdominis plane blocks: a blinded, randomized non-inferiority trial. Surg Endosc. 2020 Jul;34(7):3011-3019. doi: 10.1007/s00464-019-07097-y. Epub 2019 Sep 4. PMID 31485929